CLINICAL TRIAL: NCT00285558
Title: Peer-Enhanced Intervention to Support Teen Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK62916 (completed); R01DK062916 (NIH)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: obesity; adolescent; weight loss; body mass index; evaluation studies; peer group; behavior therapy; diet; exercise; self efficacy; parents
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

ARMS (2):
- CBT with peer-enhanced activities (Experimental): Cognitive behavioral treatment (CBT) with peer-enhanced adventure therapy. The peer intervention, ''adventure therapy,'' is based on the principles of Outward Bound and was expected to affect weight status through a positive effect on self-concept.
  Interventions: Behavioral: CBT with peer-enhanced activities
- CBT with supervised aerobic exercise (Active Comparator): Cognitive behavioral treatment (CBT) with supervised aerobic exercise. Activities for the supervised exercise intervention included use of treadmills, stationary bicycles, and other aerobic activities selected by participants, including dance videos and brisk walking within the clinic setting.
  Interventions: Behavioral: CBT with supervised aerobic exercise

INTERVENTIONS:
Behavioral: CBT with peer-enhanced activities
  Arms: CBT with peer-enhanced activities
Behavioral: CBT with supervised aerobic exercise
  Arms: CBT with supervised aerobic exercise

SUMMARY:
The purpose of this study is to determine whether adding a peer-based intervention based on an outward bound model is more effective than a standard behavioral weight intervention for helping adolescents lose weight.

DETAILED DESCRIPTION:
The prevalence of overweight in children and adolescents has increased significantly during the last two decades. While there are empirically supported weight management interventions for school age children, treatment findings with overweight adolescents are not as consistent. A potential limitation of weight control interventions for adolescents is the minimal attention given to the peer group as an active component of treatment. We have promising findings from a pilot study that involves adding an innovative peer-based intervention (peer-based skills training; PBST) to cognitive- behavioral weight management treatment for adolescents. The purpose of the proposed study is to expand the pilot by: 1) increasing our sample size, 2) assessing weight loss over a longer time period, and 3) evaluating the role of psychosocial variables, as well as physical activity and diet, in mediating treatment outcome. It is hypothesized that overweight adolescents randomized to cognitive-behavioral treatment with peer enhancement will demonstrate greater weight loss at long term follow-up than adolescents randomized to cognitive-behavioral treatment with exercise.

One hundred and fifty adolescents between the ages of 13 and 16 years and 20% and 90% overweight will be randomized to one of two treatment conditions: 1) Cognitive-Behavioral Weight Loss Treatment with Peer-Based Skills Training (CBT+PBST) or 2) Cognitive-Behavioral Weight Loss Treatment with Exercise (CBT+EXER). Measures of height, weight, physical activity, diet, and psychosocial functioning will be obtained at baseline, end of treatment, 12 months, and 24 months after randomization. A between-groups t-test will be conducted to evaluate group differences in change in percent overweight between baseline and 24-month follow-up. Hierarchical linear modeling will be used to assess the pattern of weight loss for the two treatment groups across four time points: baseline, end of treatment, 12 month, and 24 month follow-up. Effects of treatment on psychosocial measures will be analyzed using mixed analysis of variance with treatment condition as the between subjects factor and a within subject factor of time. Finally, a series of regression analyses will be conducted to evaluate the role of psychosocial variables, physical activity, and diet, as mediators of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 13-16 years old
* 20-90% overweight with reference gender and age
* At least 1 parent who can participate
* English speaking
* Agree to study participation and random assignment
* Be available for long-term follow-up

Exclusion Criteria:

* Current involvement in another weight loss program
* Unable to adhere to prescribed dietary plan and physical activity due to medical condition
* Unable to understand intervention materials
* In treatment for or diagnosed with psychiatric disorder

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent Body Mass Index (BMI) | 12 and 24 months

SECONDARY OUTCOMES:
Self concept | 12 and 24 months
  Self- Perception Profile for Adolescents and the Physical Self-Worth Scale

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Jelalian, PhD, Principal Investigator — Brown University Medical School; Lifespan Corporation
Locations (1):
- Bradley Hasbro Children's Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Result] Jelalian E, Lloyd-Richardson EE, Mehlenbeck RS, Hart CN, Flynn-O'Brien K, Kaplan J, Neill M, Wing RR. Behavioral weight control treatment with supervised exercise or peer-enhanced adventure for overweight adolescents. J Pediatr. 2010 Dec;157(6):923-928.e1. doi: 10.1016/j.jpeds.2010.05.047. Epub 2010 Jul 23. PMID 20655544
- [Derived] Rancourt D, Barker DH, Jelalian E. Sex as a Moderator of Adolescents' Weight Loss Treatment Outcomes. J Adolesc Health. 2018 May;62(5):591-597. doi: 10.1016/j.jadohealth.2017.12.002. Epub 2018 Mar 7. PMID 29525290